CLINICAL TRIAL: NCT00135213
Title: PROS Brief Smoking Cessation Counseling in Pediatric Practice to Reduce Secondhand Smoke Exposure of Young Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Truth Initiative (Other); Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 11585
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2006-09

CONDITIONS: Health Care Quality, Access, and Evaluation; Smoking Cessation
Keywords: passive smoking; pediatric practice; smoking cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: training in smoking cessation

SUMMARY:
The investigators' long-term goal is to improve the quality of services targeting the prevention of secondhand smoke (SHS). Their specific aims are to:

* refine components of office systems and counseling interventions for parental tobacco control in pediatric outpatient settings; and
* pilot test the feasibility and efficacy of a parental tobacco control randomized controlled trial in pediatric office settings using 5 intervention and 5 comparison pediatric practice sites.

The investigators hypothesize that:

* clinicians in intervention practices (compared to those in control practices) will more often implement successful office systems, screen for parental smoking, advise parents to quit and to prohibit smoking and SHS exposure at home, recommend pharmacotherapy, provide adjuncts, and refer parents to cessation programs; and
* parents who smoke in intervention practices (measured by 3-month follow-up telephone surveys) will be more likely than those in control practices to have received cessation services, use pharmacotherapy, make lasting quit attempts, and institute rules to prohibit smoking and limit SHS exposure at home.

DETAILED DESCRIPTION:
The investigators' long-term goal is to improve the quality of services targeting the prevention of secondhand smoke (SHS). Their specific aims are to:

* refine components of office systems and counseling interventions for parental tobacco control in pediatric outpatient settings; and
* pilot test the feasibility and efficacy of a parental tobacco control randomized controlled trial in pediatric office settings using 5 intervention and 5 comparison pediatric practice sites.

The investigators hypothesize that:

* clinicians in intervention practices (compared to those in control practices) will more often implement successful office systems, screen for parental smoking, advise parents to quit and to prohibit smoking and SHS exposure at home, recommend pharmacotherapy, provide adjuncts, and refer parents to cessation programs; and
* parents who smoke in intervention practices (measured by 3-month follow-up telephone surveys) will be more likely than those in control practices to have received cessation services, use pharmacotherapy, make lasting quit attempts, and institute rules to prohibit smoking and limit SHS exposure at home.

ELIGIBILITY:
Inclusion Criteria:

* PROS practices will be eligible to participate if they are located in a community-based setting with a non-institutionalized population.
* Physicians are eligible if they are able and willing to provide informed consent and have a patient flow of several children per week, and are not currently participating in another PROS study. They also must be able to read and speak English.
* Eligible parents will:

  * be parents or guardians age 18 or older;
  * be parents of a child aged 0-6;
  * have access to a telephone; and
  * be able to speak/read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2005-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
rates of reduced exposure to secondhand smoke

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Klein, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States